CLINICAL TRIAL: NCT03482635
Title: A Phase II/III Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Safety and Efficacy of BI655130 (SPESOLIMAB) Induction Therapy in Patients With Moderate-to-severely Active Ulcerative Colitis Who Have Failed Previous Biologics Therapy
Brief Title: BI655130 (SPESOLIMAB) Induction Treatment in Patients With Moderate-to-severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1368-0005; 2017-004230-28 (EudraCT Number)
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Results first posted 2021-06-11 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1- Placebo Group (Experimental)
  Interventions: Drug: Placebo
- Group 2- Small Dose Group (Experimental)
  Interventions: Drug: Spesolimab
- Group 3- Medium Dose Group (Experimental)
  Interventions: Drug: Spesolimab
- Group 4 - High Dose Group (Experimental)
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — Solution for infusion
  Arms: Group 2- Small Dose Group; Group 3- Medium Dose Group; Group 4 - High Dose Group
Drug: Placebo — Solution for infusion
  Arms: Group 1- Placebo Group

SUMMARY:
This trial has two sequentially enrolling parts with different objectives. The primary objectives of this trial are

* to prove the concept of clinical activity of BI655130 (SPESOLIMAB) in patients with moderate-to-severely active ulcerative colitis who have failed previous biologic treatments and to identify efficacious and safe dose regimens in Part 1 (Phase II)
* to confirm efficacy and safety of BI655130 (SPESOLIMAB) in patients with moderate-to-severely active ulcerative colitis who have failed previous biologic treatments in Part 2 (Phase III)
* To provide, along with induction study 1368-0018 and the run-in cohort of 1368-0020, the target population to be evaluated in study 1368-0020.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years, at date of signing informed consent, males or females
* Diagnosis of ulcerative colitis ≥ 3 months prior to screening by clinical and endoscopic evidence corroborated by a histopathology report
* Moderate to severe activity (total MCS 6 to 12 with a RBS ≥ 1 AND an SFS ≥ 1 AND mESS ≥ 2 within 7-28 days prior to first dose)
* Endoscopic activity extending proximal to the rectum (≥ 15 cm from anal verge)
* Well-documented demonstration of inadequate response or loss of response or have had unacceptable side effects with approved doses of TNFɑ antagonists (infliximab, adalimumab, golimumab) and/or vedolizumab in the past (screening of both TNFɑ antagonists-AND-Vedolizumab failure patients will be capped once 48 randomized patients in Part 1 and 117 randomized patients in Part 2 meet this criterion; patients who have already been screened at the time of the cap will continue to be randomized into the study)
* Further inclusion criteria apply

Exclusion Criteria:

* Evidence of abdominal abscess at screening
* Evidence of fulminant colitis or toxic megacolon at screening
* Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine
* Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (13):
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - University of Miami, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - University of Chicago, Chicago, Illinois
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - Baylor College of Medicine, Houston, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
- Austria (2):
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern, Linz
  - AKH - Medical University of Vienna, Vienna
- Belgium (2):
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Canada (3):
  - University of Manitoba - Health Sciences Centre, Winnipeg, Manitoba
  - Victoria Hospital (LHSC), London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Germany (7):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen AöR, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Ulm, Ulm
- Italy (2):
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Istituto Clinico Humanitas, Rozzano (MI)
- Japan (9):
  - Toho University Sakura Medical Center, Chiba, Sakura
  - Sapporo Tokushukai Hospital, Hokkaido, Sapporo
  - Sapporo Higashi Tokushukai Hospital, Hokkaido, Sapporo
  - Hyogo College of Medicine Hospital, Hyogo, Nishinomiya
  - Sameshima Hospital, Kagoshima, Kagoshima
  - Ofuna Chuo Hospital, Kanagawa, Kamakura
  - Tokyo Medical and Dental University, Tokyo, Bunkyo-ku
  - Kitasato Institute Hospital, Tokyo, Minato-ku
  - Tokyo Yamate Medical Center, Tokyo, Shinjuku
- Poland (2):
  - Health Center of Mother, Child and Youth Sp.z o.o., Warsaw
  - Central Clinical Hospital MSWiA, Internal Diseases, Warsaw, Warsaw
- Russia (6):
  - FSB Instit. HC Irkutsk Scient.Cent. Sibirian Branch of Russ. Acad. Scien., Irkutsk
  - Kirov State Med.Univ. of MoH RF, Kirov
  - Federal State Budgetary Institution " State Scientific Center of Coloproctology" MOH Russia, Moscow
  - Reg. Clin. Scientific Research Institute na Vladimiskiy, Moscow
  - The limited liability company "Clinic USI 4D", Pyatigorsk
  - FSBMEI HPE "Military Medical Academy n.a. S.M. Kirov", Saint Petersburg
- South Korea (2):
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
- Spain (2):
  - Hospital Virgen del Rocío, Seville
  - Hospital Politècnic La Fe, Valencia
- United Kingdom (4):
  - Barnsley Hospital, Barnsley
  - Doncaster Royal Infirmary, Doncaster
  - Guy's Hospital, London
  - Whiston Hospital, Prescot

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Lebwohl MG, Thoma C, Haeufel T. Spesolimab use in generalised pustular psoriasis flares - Authors' reply. Lancet. 2024 Aug 31;404(10455):847-848. doi: 10.1016/S0140-6736(24)01557-5. No abstract available. PMID 39216969
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase II/III randomized, placebo-controlled, double-blind trial to assess the safety and efficacy of spesolimab induction therapy in patients with moderate-to-severely active ulcerative colitis who have failed previous biologics therapy. Phase III was not conducted, due to recruitment issues in Phase II.
Pre-assignment Details: Only subjects that met all the study inclusion and non of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue medication was allowed for all patients as required.
Groups:
- Placebo: A solution of placebo was administered as intravenous infusion once every 4 weeks over a period of 12 weeks, (at week 0, week 4, week 8) in patients with moderate to severe ulcerative colitis who had failed previous biological treatments in the past.
- 300 mg Spesolimab (BI 655130) SD: A single dose (SD) of 300 milligram (mg) solution of spesolimab was administered as intravenous infusion at week 0 in patients with moderate to severe ulcerative colitis who had failed previous biological treatments in the past.
- 450 mg Spesolimab (BI 655130) q4w: 450 mg solution of spesolimab was administered, as intravenous infusion, once every 4 weeks (q4w) over a period of 12 weeks, (at week 0, week 4, week 8) in patients with moderate to severe ulcerative colitis who had failed previous biological treatments in the past.
- 1200 mg Spesolimab (BI 655130) q4w: 1200 mg solution of spesolimab was administered, as intravenous infusion, once every 4 weeks (q4w) over a period of 12 weeks, (at week 0, week 4, week 8) in patients with moderate to severe ulcerative colitis who had failed previous biological treatments in the past.
Period: Overall Study
Arm/Group | Placebo | 300 mg Spesolimab (BI 655130) SD | 450 mg Spesolimab (BI 655130) q4w | 1200 mg Spesolimab (BI 655130) q4w
Started | 23 | 24 | 23 | 28
Treated | 23 | 24 | 23 | 27
Completed (Completed trial medication) | 18 | 21 | 22 | 20
Not Completed | 5 | 3 | 1 | 8
Not completed — Lack of Efficacy | 0 | 0 | 1 | 3
Not completed — Adverse Event | 2 | 2 | 0 | 3
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 1
Not completed — Withdrawn by Principle Investigator | 1 | 0 | 0 | 0
Not completed — Not treated | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomised Set: The RS included all randomised patients. Treatment assignment was as randomised. It was the main analysis set for presentation of efficacy on binary endpoints.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 300 mg Spesolimab (BI 655130) SD | 450 mg Spesolimab (BI 655130) q4w | 1200 mg Spesolimab (BI 655130) q4w | Total
Number analyzed (Participants) | 23 | 24 | 23 | 28 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (14.1) | 41.4 (14.6) | 42.3 (15.3) | 43.9 (14.9) | 42.5 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 10 | 8 | 36
  Male | 12 | 17 | 13 | 20 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 23 | 24 | 23 | 27 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 4 | 1 | 4 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 18 | 23 | 18 | 21 | 80
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Clinical Remission at Week 12
Description: Proportion of patients with clinical remission (defined as modified Mayo Clinical Score (MCS) ≤ 2, with Stool Frequency Score (SFS) = 0 or 1 [if drop ≥1 from baseline] and Rectal Bleeding Score (RBS) = 0 and modified Endoscopic Subscore (mESS) ≤ 1) at week 12.
  Proportion of patients was calculated as n/N, with n=number of patients with clinical remission at week 12 and N=number analyzed. 95% Confidence Intervals (CI) were calculated using the method of Wilson.
Time Frame: At week 12.
Population: Randomised Set - Non Response Imputation (RS-NRI): The randomised set included all randomised patients, including patients with non-response imputation.
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Placebo | 300 mg Spesolimab (BI 655130) SD | 450 mg Spesolimab (BI 655130) q4w | 1200 mg Spesolimab (BI 655130) q4w
Number analyzed (Participants) | 23 | 24 | 23 | 28
Proportion of Participants | 0.00 [0.000 to 0.143] | 0.042 [0.007 to 0.202] | 0.087 [0.024 to 0.268] | 0.071 [0.020 to 0.226]
Statistical Analysis 1: Comparison: Placebo vs 300 mg Spesolimab (BI 655130) SD; Test type: Other; Risk Difference (RD) = 0.042, 95% CI 2-sided [-0.105 to 0.202] — Unadjusted absolute risk difference to placebo, [Treatment - Placebo]. 95% CI for risk difference were calculated using the method of Newcombe
Statistical Analysis 2: Comparison: Placebo vs 450 mg Spesolimab (BI 655130) q4w; Test type: Other; Risk Difference (RD) = 0.087, 95% CI 2-sided [-0.069 to 0.268] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs 1200 mg Spesolimab (BI 655130) q4w; Test type: Other; Risk Difference (RD) = 0.071, 95% CI 2-sided [-0.081 to 0.226] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Proportion of Patients With Clinical Response at Week 12
Description: Proportion of patients with clinical response (defined as Rectal Bleeding Score (RBS) ≤ 1 or decrease by ≥1 from baseline; and total Mayo Clinical Score (MCS) decrease by ≥ 3 and 30% from baseline) at week 12. Proportion of patients is calculated as n/N, with n=number of patients with clinical response at week 12 and N=number of patients analyzed. 95% Confidence Intervals (CI) are calculated using the method of Wilson.
Time Frame: At week 12.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | 300 mg Spesolimab (BI 655130) SD | 450 mg Spesolimab (BI 655130) q4w | 1200 mg Spesolimab (BI 655130) q4w
Number analyzed (Participants) | 23 | 24 | 23 | 28
Proportion of participants | 0.217 [0.097 to 0.419] | 0.167 [0.067 to 0.359] | 0.261 [0.125 to 0.465] | 0.250 [0.127 to 0.434]
Statistical Analysis 1: Comparison: Placebo vs 300 mg Spesolimab (BI 655130) SD; Test type: Other; Risk Difference (RD) = -0.051, 95% CI 2-sided [-0.276 to 0.176] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 450 mg Spesolimab (BI 655130) q4w; Test type: Other; Risk Difference (RD) = 0.043, 95% CI 2-sided [-0.199 to 0.280] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs 1200 mg Spesolimab (BI 655130) q4w; Test type: Other; Risk Difference (RD) = 0.033, 95% CI 2-sided [-0.204 to 0.252] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Proportion of Patients With Endoscopic Improvement at Week 12
Description: Proportion of patients with endoscopic improvement at week 12 (defined as modified Endoscopic Subscore (mESS) ≤ 1) Proportion of patients was calculated as n/N, with n=number of patients with Endoscopic Improvment at Week 12 and N=number analysed. 95% Confidence Intervals (CI) were calculated using the method of Wilson.
Time Frame: At week 12.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | 300 mg Spesolimab (BI 655130) SD | 450 mg Spesolimab (BI 655130) q4w | 1200 mg Spesolimab (BI 655130) q4w
Number analyzed (Participants) | 23 | 24 | 23 | 28
Proportion of participants | 0.000 [0.000 to 0.143] | 0.083 [0.023 to 0.258] | 0.087 [0.024 to 0.268] | 0.071 [0.020 to 0.226]
Statistical Analysis 1: Comparison: Placebo vs 300 mg Spesolimab (BI 655130) SD; Test type: Other; Risk Difference (RD) = 0.083, 95% CI 2-sided [-0.072 to 0.258] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs 450 mg Spesolimab (BI 655130) q4w; Test type: Other; Risk Difference (RD) = 0.087, 95% CI 2-sided [-0.069 to 0.268] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs 1200 mg Spesolimab (BI 655130) q4w; Test type: Other; Risk Difference (RD) = 0.071, 95% CI 2-sided [-0.081 to 0.226] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Proportion of Patients With Combined Endoscopic Improvement and Histologic Remission at Week 12
Description: Proportion of patients with combined endoscopic improvement and histologic remission at week 12 (defined as modified Endoscopic Subscore (mESS) ≤ 1 and Robarts Histology Index ≤ 6). Proportion of patients was calculated as n/N, with n= number of patients with Endoscopic Improvement and histologic remission at week 12 and N=number of patients analysed.
Time Frame: At week 12.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | 300 mg Spesolimab (BI 655130) SD | 450 mg Spesolimab (BI 655130) q4w | 1200 mg Spesolimab (BI 655130) q4w
Number analyzed (Participants) | 23 | 24 | 23 | 28
Proportion of participants | 0.00 [0.000 to 0.143] | 0.083 [0.023 to 0.258] | 0.043 [0.008 to 0.210] | 0.036 [0.006 to 0.177]
Statistical Analysis 1: Comparison: Placebo vs 300 mg Spesolimab (BI 655130) SD; Test type: Other; Risk Difference (RD) = 0.083, 95% CI 2-sided [-0.072 to 0.258] — Unadjusted absolute risk difference to placebo, [Treatment - Placebo]
Statistical Analysis 2: Comparison: Placebo vs 450 mg Spesolimab (BI 655130) q4w; Test type: Other; Risk Difference (RD) = 0.043, 95% CI 2-sided [-0.104 to 0.210] — Unadjusted absolute risk difference to placebo, [Treatment - Placebo]
Statistical Analysis 3: Comparison: Placebo vs 1200 mg Spesolimab (BI 655130) q4w; Test type: Other; Risk Difference (RD) = 0.036, 95% CI 2-sided [-0.110 to 0.177] — Unadjusted absolute risk difference to placebo, [Treatment - Placebo]

5. Secondary Outcome: Change in Inflammatory Bowel Disease Questionnaire (IBDQ) Score From Baseline at Week 12
Description: Change in Inflammatory Bowel Disease Questionnaire (IBDQ) score from baseline at Week 12.
  The IBDQ is a 32-item self-report questionnaire for patients with IBD to evaluate the patient reported outcomes across 4 dimensions: bowel symptoms (loose stools, abdominal pain), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). The response options describe the magnitude or frequency of impairment from 1 (most severe) to 7 (no impairment). The items are summed up, resulting in a sum score ranging from 32 to 224 points, with higher scores indicating better outcomes. A score change of 16 is reported to reflect the minimal clinically important difference (MCID).
  Mean is adjusted mean.
Time Frame: At baseline and at week 12.
Population: Modified Randomised Set (m-RS): The m-RS included all patients in the RS who had a baseline and at least 1 post-baseline measurement for the endpoint under consideration. Treatment assignment was randomised.
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Placebo | 300 mg Spesolimab (BI 655130) SD | 450 mg Spesolimab (BI 655130) q4w | 1200 mg Spesolimab (BI 655130) q4w
Number analyzed (Participants) | 18 | 19 | 21 | 18
Score on a scale | 19.8 [4.7 to 35.0] | 19.5 [4.6 to 34.5] | 21.2 [6.6 to 35.9] | 20.8 [6.3 to 35.4]
Statistical Analysis 1: Comparison: Placebo vs 300 mg Spesolimab (BI 655130) SD; Restricted maximum likelihood (REML)-based repeated measures approach. The model included fixed, categorical effects of treatment, visit, and treatment by visit interaction, and stratification factors (prior biologic treatment failure and concomitant corticosteroid therapy at Visit 2/randomisation), as well as the continuous fixed covariates of baseline and baseline-by-visit interaction. An unstructured covariance structure was used to model the within-patient measurements; Test type: Other; p = 0.9776, Mixed Models Analysis; Difference of adjusted means = -0.3, 95% CI 2-sided [-21.6 to 21.0], Standard Error of Mean 10.7
Statistical Analysis 2: Comparison: Placebo vs 450 mg Spesolimab (BI 655130) q4w; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.8940, Mixed Models Analysis; Difference of adjusted means = 1.4, 95% CI 2-sided [-19.6 to 22.4], Standard Error of Mean 10.6
Statistical Analysis 3: Comparison: Placebo vs 1200 mg Spesolimab (BI 655130) q4w; [analysis description as in outcome 5, analysis 1]; Test type: Other; p = 0.9241, Mixed Models Analysis; Difference of adjusted means = 1.0, 95% CI 2-sided [-20.0 to 22.1], Standard Error of Mean 10.6

ADVERSE EVENTS:
Time Frame: From screening until end of study, up to 29 weeks.
Description: Safety Analysis Set (SAF): All patients who were randomised and received at least one dose of study drug.
Arm/Group | Placebo | 300 mg Spesolimab (BI 655130) SD | 450 mg Spesolimab (BI 655130) q4w | 1200 mg Spesolimab (BI 655130) q4w
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24 | 0/23 | 0/27
Serious Adverse Events (participants affected / at risk) | 4/23 | 3/24 | 2/23 | 3/27
Other Adverse Events (participants affected / at risk) | 5/23 | 7/24 | 7/23 | 17/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | 300 mg Spesolimab (BI 655130) SD (N=24) | 450 mg Spesolimab (BI 655130) q4w (N=23) | 1200 mg Spesolimab (BI 655130) q4w (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | 300 mg Spesolimab (BI 655130) SD (N=24) | 450 mg Spesolimab (BI 655130) q4w (N=23) | 1200 mg Spesolimab (BI 655130) q4w (N=27)
Anaemia (Blood and lymphatic system disorders) | 5 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 2 | 1 | 6
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 2
Feeling hot (General disorders) | 0 | 0 | 3 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 3
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2

LIMITATIONS AND CAVEATS:
Due to recruitment issues during phase II, the trial was prematurely ended according to a protocol defined option. Phase III was not conducted. The trial was completed as defined in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation of review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT03482635/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/35/NCT03482635/SAP_001.pdf